CLINICAL TRIAL: NCT01268189
Title: Evaluation of Oxygen Diffusion Dressing for Accelerating Healing of Donor Site and Other Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-09-008
Record Dates: First submitted 2010-12-21; First posted 2010-12-29 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Burns
Keywords: burn wound; management with oxygen
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Burn wound patients with donor sites (Experimental): Oxygen diffusing dressing applied to wound vs standard of care dressing (Xeroform) applied to wound (patient serves as own control as s/he receives 1 dressing on 1 donor site and the other on a 2nd donor site)
  Interventions: Device: Oxygen diffusing dressing; Device: Standard of care dressing

INTERVENTIONS:
Device: Oxygen diffusing dressing — Oxygen diffusing dressing applied to study wound
  Other Names: OxyBand dressing
Device: Standard of care dressing — Xeroform control dressing applied to control wound
  Other Names: Xeroform dressing

SUMMARY:
This is a single-center, prospective, randomized, and controlled study to evaluate the effectiveness of OxyBand Dressing for the use as a dressing for autogenous skin donor sites compared to our current standard donor site dressing (Xeroform). Hypothesis is that the mean healing time for wounds treated with the OxyBand dressing will be less than the mean healing time for wounds treated with the Xeroform dressing.

DETAILED DESCRIPTION:
Patients who are scheduled for excision of burns or other injuries will have one of two donor sites covered with the OxyBand Dressing, and the other treated according to standard of care. OxyBand is an FDA (Food and Drug Administration) approved (K043063) wound dressing for delivery of oxygen into the wound. Two small clinical studies using OxyBand have been conducted on standardized laser burn wounds, demonstrating faster healing time compared to a placebo. No studies have compared this dressing to Xeroform dressing, the standard dressing used on donor sites in the USAISR.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age; of either gender and in good general health.
* Subject has sustained burn wounds of less than 30 percent of the total body surface area
* Burn wounds do not involve the harvesting area
* Subject has sustained burn wounds that, in the judgment of the attending surgeon, require excision and grafting of sufficient extent to justify two donor sites of equal and symmetrical size on non-dependent body surfaces areas
* The scheduled excision and grafting procedure is the first such operation for the subject during this hospitalization
* Subject agrees to participate in follow-up evaluations

Exclusion Criteria:

* Critical illnesses such as those requiring ventilator support, or having a systemic infection or hemodynamic instability, defined as a mean arterial pressure less than 60 or requiring vasoactive medications to support blood pressure
* Major acute or chronic medical illnesses that could affect wound healing (e.g. peripheral vascular disease, insulin dependent diabetes, blood clotting disorder)
* Subjects receiving treatment with medications that inhibit or compromise wound healing. Examples include therapeutic anticoagulants, antiplatelet drugs, and systemic steroids such as warfarin, clopidogrel or prednisone. The use of anticoagulants does not include DVT (Deep Vein Thrombosis) prophylaxis. Subjects may use aspirin or lovenox
* Cellulitis or other infection of the potential donor sites
* Donor site has been previously harvested for grafting
* Subjects with greater than 30% total body surface area burns
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly F Lairet, MD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Burn Center, Fort Sam Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Burn Wound Patients: Burn wound patients with experimental (oxyband) and control (Xeroform) dressings placed on 2 separate skin graft donor sites
Period: Overall Study
Arm/Group | Burn Wound Patients
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Subjects serve as their own control as experimental and standard of care dressings applied to 2 different donor sites. Total of 17 participants completed, with 34 donor sites.
Groups:
- Burn Wound Patients: Burn wound patients with oxygen diffusing dressing placed on 1 donor skin graft site and standard of care (Xeroform) dressing placed on a 2nd donor skin graft
Arm/Group | Burn Wound Patients
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 35 [20 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Burn Size [Mean (Full Range); unit: percentage of total skin area] | 9.2 [2 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Healing Time for Donor Site Wounds
Description: Wounds are inspected on postoperative days 4, 8, and then every two days until the wound is deemed to be healed.
Time Frame: number of days to healing
Measure: Mean (Standard Deviation); unit: days
Groups:
- Study Dressing: Oxygen diffusing dressing applied to wound
  Oxygen diffusing dressing: Oxygen diffusing dressing applied to study wound
- Control Dressing: Xeroform (current standard of care) dressing applied to wound
  Control dressing: Xeroform control dressing applied to control wound
Arm/Group | Study Dressing | Control Dressing
Number analyzed (Participants) | 17 | 17
days | 9.4 (1.7) | 12.4 (2.7)

2. Secondary Outcome: Pain Perceived by Patient
Description: Patient will be asked to rate pain 0-10 (0=no pain, 10=maximum pain) at the study site and the control site. Used Visual Analogue Scale (VAS) for this purpose.
Time Frame: Post-Operative Day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Dressing | Control Dressing
Number analyzed (Participants) | 17 | 17
units on a scale | 0.6 (1.6) | 1.6 (1.9)

3. Secondary Outcome: Patient Will be Asked to Rate Pain 0-10/10 at the Study Site and the Control Site
Time Frame: Post-Operative Day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Dressing | Control Dressing
Number analyzed (Participants) | 17 | 17
units on a scale | 0.4 (1.3) | 1.4 (2.2)

4. Secondary Outcome: Patient Will be Asked to Rate Pain 0-10/10 at the Study Site and the Control Site
Time Frame: Post-Operative Day 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Dressing | Control Dressing
Number analyzed (Participants) | 17 | 17
units on a scale | 0.3 (1) | 0.8 (1.5)

5. Secondary Outcome: Patient Will be Asked to Rate Pain 0-10/10 at the Study Site and the Control Site
Time Frame: Post-Operative Day 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Dressing | Control Dressing
Number analyzed (Participants) | 17 | 17
units on a scale | 0.2 (0.8) | 0.5 (1.2)

ADVERSE EVENTS:
Arm/Group | Study Dressing | Control Dressing
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Dressing (N=17) | Control Dressing (N=17)
Blistering (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes